CLINICAL TRIAL: NCT01547208
Title: Does Timing of VT Ablation Affect Prognosis in Patients With an Implantable Cardioverter-defibrillator?
Acronym: PARTITA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Paolo Della Bella, Director of Arrhythmia Department and Clinical Electrophysiology Laboratories, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PARTITA
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Ventricular Tachycardias
Keywords: ICD shocks; Ventricular tachycardias ablation; Timing of ablation; Electrical storm; Arrhythmic storm
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Patients will be randomized to a VT ablation procedure immediately after an appropriate ICD shock
  Interventions: Procedure: Immediate radiofrequency ablation of ventricular tachycardia
- Group B (Active Comparator): Patients will wait until an arrhythmic storm to undergo a VT ablation procedure
  Interventions: Procedure: Radiofrequency ablation of ventricular tachycardia

INTERVENTIONS:
Procedure: Immediate radiofrequency ablation of ventricular tachycardia — Radiofrequency ablation of ventricular tachycardia is performed immediately after an appropriate ICD shock
  Arms: Group A
Procedure: Radiofrequency ablation of ventricular tachycardia — Radiofrequency ablation of ventricular tachycardia will be performed after an arrhythmic storm occurs
  Arms: Group B

SUMMARY:
The purpose of this study is to assess whether the burden of untreated non-sustained ventricular tachycardias (VTs), or episodes treated with anti-tachycardia pacing, correlates with appropriate implantable cardiac defibrillator (ICD) shock therapies and to evaluate if the timing of radiofrequency VT ablation affects the prognosis of ICD recipients.

DETAILED DESCRIPTION:
Enrolled patients will remain in a first phase of the study until the first appropriate ICD shock will be delivered.

The objective of this first stage is to assess whether the burden of untreated non sustained VTs or episodes treated with anti-tachycardia pacing is predictive of appropriate ICD shocks.

The second phase of the study will start after the first appropriate ICD shock delivered for VT.

Patients will be then randomized to immediate VT ablation or to standard treatment, meaning waiting until next arrhythmic storm to perform a VT ablation procedure.

The objective of this phase is compare the rate of worsening heart failure hospitalizations and deaths from any cause between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients already implanted with ICD (single-/dual -chamber, with or without cardiac resynchronization therapy) for primary or secondary prevention of sudden cardiac death

Exclusion Criteria:

Phase A exclusion Criteria:

* General contraindication to transcatheter ablation
* Contraindication to antithrombotic therapy
* Patients chronically treated with class I and III antiarrhythmic drugs

Phase B exclusion criteria:

* Patients developing first occurrence of incessant VTs
* Patients receiving a shock for first occurrence of clinically verified ventricular fibrillation
* Patients with aetiology differing from ischemic heart disease for coronary artery disease and from non-ischemic dilatative cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2012-09; Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of the first appropriate ICD shock during phase A | Event Driven
Number of patients showing worsening heart failure hospitalizations or deaths from any cause during phase B | Two Years

SECONDARY OUTCOMES:
Number of patients showing cardiac deaths during phase B | Two Years
Number of patients showing electrical storm (ES) recurrences during phase B | Two Years
Number of patients showing VT recurrences during phase B | Two Years

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Della Bella, Study Director — IRCCS San Raffaele; Andrea Radinovic, Study Director — IRCCS San Raffaele
Locations (21):
- Brussels Heart Center, Brussels, Belgium
- IKEM Hospital, Prague, Czechia
- Hôpital cardiologique du Haut-Lévêque, Bordeaux, France
- Herz und Gefass Klinik, Bad Neustadt an der Saale, Germany
- Italy (15):
  - Ospedale di Desio, Desio, Milan
  - Ospedale di Montebelluna, Montebelluna, Treviso
  - Ospedale Mater Domini, Castellanza, Varese
  - Azienda Ospedaliera Sant'Antonio Abate, Gallarate, Varese
  - Ospedale di Mirano, Mirano, Venice
  - Ospedale S. Donato, Arezzo
  - AO Policlinico di Bari, Bari
  - Ospedale Brotzu, Cagliari
  - Osp. Fondazione Giovanni Paolo II, Campobasso
  - AO Pugliese Ciaccio, Catanzaro
  - IRCCS San Raffaele, Milan
  - Fondazione G. Monasterio, Pisa
  - Policlinico Casilino, Rome
  - Azienda Ospedaliera Valtellina e Valchiavenna, Sondrio
  - Ospedale Civile Maggiore, Verona
- Centro Hospitalar Lisboa Norte, Hospital Universitário de Santa Maria, Lisbon, Portugal
- Lausanne Hospital, Lausanne, Switzerland

REFERENCES:
- [Background] Reddy VY, Reynolds MR, Neuzil P, Richardson AW, Taborsky M, Jongnarangsin K, Kralovec S, Sediva L, Ruskin JN, Josephson ME. Prophylactic catheter ablation for the prevention of defibrillator therapy. N Engl J Med. 2007 Dec 27;357(26):2657-65. doi: 10.1056/NEJMoa065457. PMID 18160685
- [Background] Kuck KH, Schaumann A, Eckardt L, Willems S, Ventura R, Delacretaz E, Pitschner HF, Kautzner J, Schumacher B, Hansen PS; VTACH study group. Catheter ablation of stable ventricular tachycardia before defibrillator implantation in patients with coronary heart disease (VTACH): a multicentre randomised controlled trial. Lancet. 2010 Jan 2;375(9708):31-40. doi: 10.1016/S0140-6736(09)61755-4. PMID 20109864
- [Background] Sweeney MO, Sherfesee L, DeGroot PJ, Wathen MS, Wilkoff BL. Differences in effects of electrical therapy type for ventricular arrhythmias on mortality in implantable cardioverter-defibrillator patients. Heart Rhythm. 2010 Mar;7(3):353-60. doi: 10.1016/j.hrthm.2009.11.027. Epub 2009 Dec 2. PMID 20185109
- [Background] Poole JE, Johnson GW, Hellkamp AS, Anderson J, Callans DJ, Raitt MH, Reddy RK, Marchlinski FE, Yee R, Guarnieri T, Talajic M, Wilber DJ, Fishbein DP, Packer DL, Mark DB, Lee KL, Bardy GH. Prognostic importance of defibrillator shocks in patients with heart failure. N Engl J Med. 2008 Sep 4;359(10):1009-17. doi: 10.1056/NEJMoa071098. PMID 18768944
- [Background] Varma N, Epstein AE, Irimpen A, Schweikert R, Love C; TRUST Investigators. Efficacy and safety of automatic remote monitoring for implantable cardioverter-defibrillator follow-up: the Lumos-T Safely Reduces Routine Office Device Follow-up (TRUST) trial. Circulation. 2010 Jul 27;122(4):325-32. doi: 10.1161/CIRCULATIONAHA.110.937409. Epub 2010 Jul 12. PMID 20625110
- [Background] Varma N, Michalski J, Epstein AE, Schweikert R. Automatic remote monitoring of implantable cardioverter-defibrillator lead and generator performance: the Lumos-T Safely RedUceS RouTine Office Device Follow-Up (TRUST) trial. Circ Arrhythm Electrophysiol. 2010 Oct;3(5):428-36. doi: 10.1161/CIRCEP.110.951962. Epub 2010 Aug 17. PMID 20716717
- [Background] Gilliam FR, Hayes DL, Boehmer JP, Day J, Heidenreich PA, Seth M, Jones PW, Stein KM, Saxon LA. Real world evaluation of dual-zone ICD and CRT-D programming compared to single-zone programming: the ALTITUDE REDUCES study. J Cardiovasc Electrophysiol. 2011 Sep;22(9):1023-9. doi: 10.1111/j.1540-8167.2011.02086.x. Epub 2011 May 31. PMID 21627705
- [Background] Carbucicchio C, Santamaria M, Trevisi N, Maccabelli G, Giraldi F, Fassini G, Riva S, Moltrasio M, Cireddu M, Veglia F, Della Bella P. Catheter ablation for the treatment of electrical storm in patients with implantable cardioverter-defibrillators: short- and long-term outcomes in a prospective single-center study. Circulation. 2008 Jan 29;117(4):462-9. doi: 10.1161/CIRCULATIONAHA.106.686534. Epub 2008 Jan 2. PMID 18172038
- [Background] Della Bella P, Baratto F, Tsiachris D, Trevisi N, Vergara P, Bisceglia C, Petracca F, Carbucicchio C, Benussi S, Maisano F, Alfieri O, Pappalardo F, Zangrillo A, Maccabelli G. Management of ventricular tachycardia in the setting of a dedicated unit for the treatment of complex ventricular arrhythmias: long-term outcome after ablation. Circulation. 2013 Apr 2;127(13):1359-68. doi: 10.1161/CIRCULATIONAHA.112.000872. Epub 2013 Feb 25. PMID 23439513
- [Background] Vergara P, Trevisi N, Ricco A, Petracca F, Baratto F, Cireddu M, Bisceglia C, Maccabelli G, Della Bella P. Late potentials abolition as an additional technique for reduction of arrhythmia recurrence in scar related ventricular tachycardia ablation. J Cardiovasc Electrophysiol. 2012 Jun;23(6):621-7. doi: 10.1111/j.1540-8167.2011.02246.x. Epub 2012 Apr 4. PMID 22486970
- [Derived] Della Bella P, Baratto F, Vergara P, Bertocchi P, Santamaria M, Notarstefano P, Calo L, Orsida D, Tomasi L, Piacenti M, Sangiorgio S, Pentimalli F, Pruvot E, De Sousa J, Sacher F, Tritto M, Rebellato L, Deneke T, Romano SA, Nesti M, Gargaro A, Giacopelli D, Peretto G, Radinovic A. Does Timing of Ventricular Tachycardia Ablation Affect Prognosis in Patients With an Implantable Cardioverter Defibrillator? Results From the Multicenter Randomized PARTITA Trial. Circulation. 2022 Jun 21;145(25):1829-1838. doi: 10.1161/CIRCULATIONAHA.122.059598. Epub 2022 Apr 3. PMID 35369700
- [Derived] Kheiri B, Barbarawi M, Zayed Y, Hicks M, Osman M, Rashdan L, Kyi HH, Bachuwa G, Hassan M, Stecker EC, Nazer B, Bhatt DL. Antiarrhythmic Drugs or Catheter Ablation in the Management of Ventricular Tachyarrhythmias in Patients With Implantable Cardioverter-Defibrillators: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Circ Arrhythm Electrophysiol. 2019 Nov;12(11):e007600. doi: 10.1161/CIRCEP.119.007600. Epub 2019 Nov 8. PMID 31698933